CLINICAL TRIAL: NCT07377721
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo and Pregabalin Capsule Controlled, Phase Ib Study to Evaluate the Efficacy and Safety of HRS-2129 in Chinese Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: A Study of HRS-2129 in Patients With Diabetic Peripheral Neuropathic Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2129-105
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: HRS-2129 compared with placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-2129 High Dose Group (Experimental)
  Interventions: Drug: HRS-2129 Tablets; Drug: HRS-2129 Placebo; Drug: Pregabalin Capsules Placebo
- HRS-2129 Low Dose Group (Experimental)
  Interventions: Drug: HRS-2129 Tablets; Drug: HRS-2129 Placebo; Drug: Pregabalin Capsules Placebo
- Pregabalin Group (Active Comparator)
  Interventions: Drug: HRS-2129 Placebo; Drug: Pregabalin Capsules
- Blank Preparation Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-2129 Placebo; Drug: Pregabalin Capsules Placebo

INTERVENTIONS:
Drug: HRS-2129 Tablets — HRS-2129 tablets.
  Arms: HRS-2129 High Dose Group; HRS-2129 Low Dose Group
Drug: HRS-2129 Placebo — HRS-2129 placebo.
Drug: Pregabalin Capsules — Pregabalin capsules.
  Arms: Pregabalin Group
Drug: Pregabalin Capsules Placebo — Pregabalin capsules placebo.
  Arms: Blank Preparation Placebo Group; HRS-2129 High Dose Group; HRS-2129 Low Dose Group

SUMMARY:
This study aims to investigate the efficacy and safety of HRS-2129 in Chinese diabetic peripheral neuropathic pain (DPNP) in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Males or females aged ≥18years of age inclusive.
3. Diagnosis of diabetic peripheral neuropathic pain (DPNP) and diabetic peripheral neuropathy (DPN) pain ≥ 3 months.
4. HbA1c ≤ 9.0% at screening and on a stable antidiabetic medication regimen for at least 30 days prior to screening as far as possible.
5. At Screening, pain scale (Visual Analog Scale, VAS) of ≥ 40 mm and < 90 mm.

Exclusion Criteria:

1. Subjects with a history of severe allergies.
2. Peripheral neuropathy or pain unrelated to diabetic peripheral neuropathy (DPN) that may confuse the assessment of diabetic peripheral neuropathic pain (DPNP).
3. Subjects with abnormal liver and renal function.
4. Corrected QT Interval (QTc): > 450 ms (male), > 470 ms (female).
5. Failure to response to previous treatment with pregabalin at doses ≥ 300 mg/d or gabapentin at doses ≥ 1200 mg/d for treatment of diabetic peripheral neuropathic pain (DPNP).
6. History of suicidal behavior or attempted suicide.
7. Participated in another clinical study within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Compare the change from baseline in Average Daily Pain Score (ADPS) between HRS-2129 and placebo at Week 4. | Baseline and Week 4.
  The mean change in Average Daily Pain Score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]). The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries.

SECONDARY OUTCOMES:
Compare the response rate between HRS-2129 and placebo at Week 4 (Proportion of subjects whose ADPS decreased by ≥ 30% and ≥ 50% from baseline). | Baseline and Week 4.
  Ratio of participants responding to treatment, as measured by Average Daily Pain Score (ADPS) reduction from baseline. The ADPS is used to determine categorical response rates.
Compare the change from baseline in ADPS between HRS-2129 and placebo at Week 1 to 4. | From Week 1 to Week 4.
  The mean change in Average Daily Pain Score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]). The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries.
Compare the change from baseline in Visual Analog Scale (VAS) between HRS-2129 and placebo at Week 4. | Baseline and Week 4.
  VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain.
Compare the change from baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) between HRS-2129 and placebo at Week 4. | Baseline and Week 4.
  Participants rate their pain in three parts of the questionnaire, which are combined into a single pain intensity score: Part 1 - 11 descriptors of pain intensity, and 4 descriptors of emotions, on a scale of 0 (none) to 3 (severe); Part 2 - a Visual Analog Scale (VAS), in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain; Part 3 - a Present Pain Intensity index in which the participant rates present pain intensity on a scale of 0 (no pain) to 5 (most intense pain).
Compare the Patient Global Impression of Change (PGIC) between HRS-2129 and placebo at Week 4. | At Week 4.
  Patient Global Impression of Change (PGIC) on a 7-point categorical scale, where 1 = very much improved and 7 = very much worse.
Compare the change from baseline in Average Daily Sleep Interference score (ADSIS) between HRS-2129 and placebo at Week 4. | Baseline and Week 4.
  The sleep interference scores on a scale of 0-10, where 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. The weekly ADSIS is based on participants daily sleep interference scores.
Number and severity of serious adverse events (SAEs). | From Week 1 to Week 6.
  To evaluate the safety of HRS-2129 during the trial.
Number and severity of adverse events (AEs). | From Week 1 to Week 6.
  To evaluate the safety of HRS-2129 during the trial.
Population Pharmacokinetics (PopPK) characteristics of HRS-2129 in Chinese patients with diabetic peripheral neuropathic pain - Serum concentration of HRS-2129. | From Day 0 to Day 30.
  Population Pharmacokinetics (PopPK) will be determined by measuring serum concentration of HRS-2129.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: Undecided